CLINICAL TRIAL: NCT06189508
Title: An Open-Label, Parallel-Group Phase I Study to Evaluate the Relative and Absolute Bioavailability of Single Subcutaneous Doses of NXT007 Among Injection Sites Abdomen, Upper Arm, and Thigh in Healthy Male Participants
Brief Title: A Study to Evaluate Single Subcutaneous Doses of NXT007 Among Injection Sites Abdomen, Upper Arm, and Thigh in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BP45057
Record Dates: First submitted 2023-12-11; First posted 2024-01-03 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Healthy Male Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: Single NXT007 SC Injection Into Abdomen (Experimental)
  Interventions: Drug: NXT007
- B: Single NXT007 SC Injection Into Upper Arm (Experimental)
  Interventions: Drug: NXT007
- C: Single NXT007 SC Injection Into Thigh (Experimental)
  Interventions: Drug: NXT007
- D: Single NXT007 IV Infusion (Experimental)
  Interventions: Drug: NXT007

INTERVENTIONS:
Drug: NXT007 — In all groups, the NXT007 single dose administration will occur in the morning of Day 1 under fasted conditions. Study treatment will occur via the route of administration and at the site of injection specified for each group.
  Other Names: RO7589655

SUMMARY:
This is a Phase I, open-label, non-randomized, parallel-group, single-dose study in healthy adult male participants. The aim is to investigate the relative bioavailability (rBA) of NXT007 among subcutaneous (SC) injection sites (abdomen, upper arm, and thigh) and the absolute bioavailability (aBA) of SC NXT007 administration. In addition, the pharmacodynamic, safety, tolerability, and immunogenicity of a single dose of NXT007 following SC or intravenous (IV) administration are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy as determined by medical evaluation that includes medical history, physical examination, vital signs, laboratory tests, and 12-lead ECG
* Body mass index (BMI) within the range of 18.5 to 30.0 kg/m^2
* Agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agree to refrain from donating sperm

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, immunological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data
* History of allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies; or known hypersensitivity to any constituent of the product
* Clinically relevant medical history and/or family history or signs of thromboembolic disease such as deep vein thrombosis
* FVIII activity ≥120 International Units per decilitre (IU/dL) at screening
* Clinically significant abnormality on electrocardiogram (ECG) at screening such as QTcF after 10-minute supine rest >450 milliseconds (ms); marked resting bradycardia (mean heart rate <40 beats per minute [bpm]); marked resting tachycardia (mean heart rate >100 bpm); or any other clinically significant ECG abnormality
* Supine systolic blood pressure at screening ≥140 millimetres of mercury (mm Hg) or <90 mm Hg or supine diastolic blood pressure at screening ≥90 mm Hg or <40 mm Hg
* Clinically significant abnormality on protein C activity (chromogenic assay), activated protein C resistance test, protein S free antigen, and/or antithrombin III activity levels
* Poor peripheral venous access
* Any other reason that, in the judgment of the investigator, would render the participants unsuitable for study participation

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) of NXT007 | At prespecified timepoints from Day 1 until Day 253
Maximum Observed Plasma Concentration (Cmax) of NXT007 | At prespecified timepoints from Day 1 until Day 253

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve up to the Last Measurable Concentration (AUC0-last) of NXT007 | At prespecified timepoints from Day 1 until Day 253
Time to Maximum Observed Plasma Concentration (tmax) of NXT007 | At prespecified timepoints from Day 1 until Day 253
Apparent Terminal Half-Life (t1/2) of NXT007 | At prespecified timepoints from Day 1 until Day 253
Apparent Clearance (CL/F) of NXT007 SC Administration | At prespecified timepoints from Day 1 until Day 253
Total Body Clearance (CL) of NXT007 IV Administration | At prespecified timepoints from Day 1 until Day 253
Volume of Distribution at Steady State of NXT007 IV Administration | At prespecified timepoints from Day 1 until Day 253
Incidence and Severity of Adverse Events | From the single dose of study treatment (Day 1) until study completion (Day 253)
Number of Participants with Abnormal Laboratory Values in Clinical Chemistry Parameters | From the single dose of study treatment (Day 1) until study completion (Day 253)
Number of Participants with Abnormal Laboratory Values in Hematology Parameters | From the single dose of study treatment (Day 1) until study completion (Day 253)
Change from Baseline in Pulse Rate at Specified Timepoints | Baseline, Days 1, 2, 3, 5, 8, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253
Change from Baseline in Tympanic Temperature at Specified Timepoints | Baseline, Days 1, 2, 3, 5, 8, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253
Change from Baseline in Systolic Blood Pressure at Specified Timepoints | Baseline, Days 1, 2, 3, 5, 8, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253
Change from Baseline in Diastolic Blood Pressure at Specified Timepoints | Baseline, Days 1, 2, 3, 5, 8, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253
Change from Baseline in Heart Rate at Specified Timepoints, as Measured by Electrocardiogram | Baseline, Days 1, 2, 8, 22, 43, 71, 141, and 253
Change from Baseline in RR, PR, QRS, QT, and QTcF Intervals at Specified Timepoints, as Measured by Electrocardiogram | Baseline, Days 1, 2, 8, 22, 43, 71, 141, and 253
Change from Baseline in Activated Partial Thromboplastin Time (aPTT) at Specified Timepoints | Baseline, Days 1, 2, 8, 15, 18, 20, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253
Change from Baseline in the Maximum Concentration of Thrombin Generated at Specified Timepoints | Baseline, Days 1, 18, 20, and 22
Prevalence of Anti-Drug Antibodies (ADAs) to NXT007 at Baseline and Incidence of ADAs to NXT007 During the Study | From Baseline until Day 253

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- New Zealand (2):
  - New Zealand Clinical Research - Auckland, Auckland
  - New Zealand Clinical Research - Christchurch, Christchurch

IPD SHARING:
Plan to Share IPD: No
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing